CLINICAL TRIAL: NCT05016791
Title: Evaluating the Impact of Prolonged, Patient-led Heart Rhythm Surveillance With the Apple Watch on Detecting Arrhythmia Recurrence and Decision-making After Catheter Ablation of Atrial Fibrillation
Brief Title: Apple Watch-led Surveillance of AF Recurrence After Catheter Ablation
Acronym: AFFU-AW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 292605
Record Dates: First submitted 2021-07-16; First posted 2021-08-23 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; wearable
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: A prospective, randomised controlled trial to compare the standard follow-up pathway after AF catheter ablation against the standard pathway augmented with Apple Watch-based rhythm monitoring. The endpoints will be the time to detection of AF recurrence and downstream sequelae such as the number of repeat ablation procedures, and longer-term freedom from AF.
Masking Description: Participants will be randomised after enrollment to active or control arms of this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Participants shall receive standard care and follow-up as provided by their clinical care provider. Heart rhythm monitoring tests shall be performed as per their clinical care provider. In addition, participants in this arm shall be loaned an Apple Watch device and undergo an education session to familiarise themselves with the study recording schedule and how to perform recordings.
  Interventions: Device: Apple Watch-based heart rhythm monitoring
- Control (No Intervention): Participants shall receive standard care and follow-up as provided by their clinical care provider. Heart rhythm monitoring tests shall be performed as per their clinical care provider.

INTERVENTIONS:
Device: Apple Watch-based heart rhythm monitoring — For the duration of the study, participants in the active arm will be asked to make ECG recordings in three circumstances:
  1. Routinely once per day from the day of randomisation till the 12-month visit after AF CA (they will be encouraged to do so at the same time each day with the option to set a reminder on the watch).
  2. If the AW requests them to do so (the automatic AF-notification algorithm will be active throughout the study period and if AF is suspected based on the tachogram, it will trigger notification for the participant to make an ECG recording). This will be till the 12-month time point.
  3. If the patient has symptoms of palpitations, pre-syncope or syncope. This will be till the 12-month time point. Monitoring should continue even if AF has been diagnosed to characterise arrhythmia burden and profile. Participants will be given the contact details of a dedicated email inbox to which to send ECGs recorded through the AW.
  Arms: Active

SUMMARY:
Atrial fibrillation (AF) is a heart rhythm disorder associated with debillitating symptoms, psychological distress and heart failure. It can also significantly increase an individuals stroke risk. Catheter ablation (CA) for AF is the most effective way to restore normal heart rhythm. However, AF can recur in up to 50% of patients after their first CA procedure and a second 'top-up' procedure may be needed to maximise effect. Early detection of recurrences can enable planning and treatment and repeat CA procedures.

Post-CA follow-up strategies rely on episodic rhythm monitoring (Holter monitor tests) that usually last between 1 and 7 days. However, AF recurrences can be intermittent and may not occur during these short monitoring episodes. A greater duration of monitoring has been shown to yield greater detection of AF recurrences.

Relying on symptoms alone to detect recurrence is also sub-optimal. AF recurrences can also be insidious. Similar symptoms may be reported from ectopy, atrial tachycardias or atrial flutter. These may require different management approaches, necessitating rhythm characterisation before considering a repeat CA.

The Apple Watch (AW) is a wristwatch that is able to monitor a wearer's heart rate and rhythm regularity as well as facilitating an immediate, real-time single-lead ECG recording. This non-invasive device that can be purchased over- the-counter has demonstrated feasibility in detecting AF and may offer a potential non-invasive, alternative long-term rhythm surveillance strategy to diagnose AF in these patients.

The investigators propose a single-centre, randomised controlled study to compare the standard follow-up strategy after index AF CA versus one supplemented with an AW-led prolonged monitoring strategy to determine if the latter will improve the expediency and rate of AF recurrence detection. Whether this will lead to improved downstream decision-making, reduction in symptomatic events and a lower prevalence of AF in the longer term will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Referred for first AFCA procedure by a Consultant electrophysiologist.
* Paroxysmal or persistent AF captured on ECG but not in continuous AF for more than 3 years. (Paroxysmal AF is defined as an episode of AF that terminates spontaneously or with intervention within 7 days of onset. Persistent AF will be defined as any continuous episode lasting longer than 7 days or requiring intervention to restore sinus rhythm after this time.)
* At least one episode of AF must have been documented by ECG or Holter within 12 months of inclusion in the study.
* Continuous anticoagulation with warfarin (INR 2-3), low molecular weight heparin, or a novel oral anticoagulant (dabigatran, apixaban, rivaroxaban, edoxaban) for ≥4 weeks prior to the ablation; or a TEE that excludes LA thrombus ≤48 hours before ablation.
* Access to a smartphone with Apple-operating system (OS) within their household for syncing with their watch.
* Participants must be able and willing to provide written informed consent

Exclusion Criteria:

* Patients with permanent AF. Permanent AF is defined as chronic, persisting AF (typically more than 1 year) for which cardioversion (pharmacologic or electrical) has failed or will never be attempted.
* Patients with AF felt to be secondary to an obvious reversible cause.
* Patients who are, or may potentially be pregnant.
* Any cardiac implantable electronic device in situ or expected to undergo implantation in the next 12 months.
* Previous left atrial (LA) ablation or LA surgery
* Pre-existing pulmonary vein stenosis or PV stent
* Pre-existing hemi-diaphragmatic paralysis
* Contraindication to anticoagulation or radiocontrast materials
* Acute coronary syndrome within 4 weeks as defined by ECG ST segment depression or prominent T-wave inversion and/or positive biomarkers of necrosis (e.g. troponin) in the absence of ST-segment elevation and in an appropriate clinical setting (chest discomfort or angina equivalent).
* Cardiac surgery, angioplasty, or cerebrovascular accident within 4 weeks prior to enrolment.
* Life expectancy less than 1 year

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Time to first documented recurrence of AF/AFl/AT | between days 91 to 365 after ablation

SECONDARY OUTCOMES:
Time to first documented recurrence of symptomatic AF/AFl/AT | between days 91 and 365 after ablation
Freedom from AF and re-do AF CA procedures per patient at the 12 month timepoint. | 1 year
The relative patient-reported satisfaction score in the active arm of the study compared to the control arm at 12 months. | 1 year
  Using the Atrial Fibrillation Quality of Life (AFeQT) survey. Min=20, Max=140. Higher score= worse outcome
The relative patient-reported satisfaction score in the active arm of the study compared to the control arm at 12 months. | 1 year
  Using the Barts Atrial Fibrillation Patient Reported Outcome Measure survey. Min=28, Max=140. Higher score= worse outcome

OTHER OUTCOMES:
Correlation between the atrial tachyarrhythmia burden during the blanking period (day 0 to day 90 post ablation) and documented recurrence of AF/AFl/AT after the blanking period ( day 91 to day 365 after ablation). | 1 year
  active arm of the study only
Per-subject comparison of accelerometer-derived activity levels during sinus rhythm as compared to atrial arrhythmia in patients who have a paroxysmal atrial arrhythmia recurrence | 1 year
  active arm of the study only

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schilling, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- St Bartholomew's Hospital, City of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No